CLINICAL TRIAL: NCT00606762
Title: A Prospective Randomized, Controlled Study Comparing Low Pressure Versus High Pressure Pneumoperitoneum During Laparoscopic Cholecystectomy.
Brief Title: Comparison Between Low Pressure Versus High Pressure Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sterling Hospital (Other)
Responsible Party: Dr. Vismit P. Joshipura, Sterling Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 1-Joshipura
Record Dates: First submitted 2008-01-22; First posted 2008-02-05 (Estimated); Last update posted 2008-02-05 (Estimated); Status verified 2008-01

CONDITIONS: Cholelithiasis
Keywords: laparoscopic cholecystectomy; low pressure pneumoperitoneum
MeSH Terms: conditions — Cholelithiasis | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- LPLC, HPLC (Active Comparator): LPLC: Low pressure pneumoperitoneum is defined as intraabdominal pressure kept at8 mm Hg after initial trocar insertion at 12 mm Hg HPLC: High pressure pneumoperitoneum is defined as intra abdominal pressure kept at 12 mm Hg throughout the procedure
  Interventions: Procedure: Laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy — Laparoscopic cholecystectomy is performed at either 8 mm Hg or 12 mm Hg intra-abdominal pressure

SUMMARY:
The physiological changes and postoperative pain are directly related with the degree of intra-abdominal pressure kept during the laparoscopy. The present study aims to examine difference between low pressure pneumoperitoneum (8 mm Hg)and High pressure pneumoperitoneum (12 mm Hg)during laparoscopic cholecystectomy in terms of pain, cardio-pulmonary function, arterial blood gas changes etc.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic gall stone disease

Exclusion Criteria:

* pyocele
* gangrene of gall bladder
* history of cholangitis
* simultaneous CBD stones
* gall stone pancreatitis
* who does not give consent if they will be randomized to LPLC

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-10; Primary Completion 2007-11 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Pain | 24 hours

SECONDARY OUTCOMES:
Pulmonary function | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Vismit P Joshipura, MS, Principal Investigator — Sterling Hospital, Ahmedabad
Locations (1):
- Sterling Hospital, Ahmedabad, Gujarat, India